CLINICAL TRIAL: NCT01055028
Title: Paclitaxel in Combination With Bevacizumab (Avastin) for the Treatment of Metastatic or Unresectable Angiosarcoma
Brief Title: Paclitaxel + Bevacizumab (Avastin) for the Treatment of Metastatic or Unresectable Angiosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Stanford University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kristen Ganjoo, Assistant Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17755; SU-01202010-4743 (Other: Stanford University); SARCOMA0006 (Other: OnCore)
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2017-05

CONDITIONS: Angiosarcomas; Soft Tissue Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma | interventions — Bevacizumab; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A / Treatment 1 (Experimental): Participants were to receive paclitaxel 200 mg/m² intravenously over 3 hours every 21 days followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3 to 6: 30 min) every 21 days x 6 cycles.
  Maintenance bevacizumab (MB), 15 mg/kg once every 21 days intravenously for a maximum of 8 cycles, was initiated after the completion of paclitaxel + bevacizumab combination.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel
- Regimen B / Treatment 2 (Experimental): Patients were to receive paclitaxel 90 mg/m² weekly x 3 of a 28-day cycle followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3 to 6: 30 min) every 21 days x 6 cycles.
  Maintenance bevacizumab (MB), 15 mg/kg once every 21 days intravenously for a maximum of 8 cycles, was initiated after the completion of paclitaxel + bevacizumab combination.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg, IV every 21 days x 6 cycles.
  Other Names: Avastin
Drug: Paclitaxel — Regimen A / Treatment 1: 200 mg/m² IV over 3 hours every 21 days.
  Regimen B / Treatment 2: 90 mg/m² weekly x 3 of a 28-day cycle
  Other Names: Abraxane

SUMMARY:
This is an open-label, single-arm, multi-center, Phase 2 study with Paclitaxel in combination with Bevacizumab in patients with Unresectable or Metastatic Angiosarcoma. The study aims to determine the safety and effectiveness of combining two drugs Paclitaxel and Bevacizumab in the treatment of Angiosarcoma that cannot be removed by surgery, or has spread to other parts of your body. The primary objective is to evaluate 4month non progression rate. The secondary objective is to evaluate overall response rate after 3rd and 6th cycle, median duration of response, 6th and 12th month survival, toxicity of Paclitaxel and Bevacizumab combination, toxicity of maintenance Bevacizumab and to collect paraffin-embedded tumor blocks for angiogenesis markers and tissue microarray.

DETAILED DESCRIPTION:
Regimen A versus B was chosen at the discretion of the treating physician. Both groups were analyzed together as far as outcome.

Patients were to receive paclitaxel 200 mg/m2 intravenously over 3 hours every 21 days (Regimen A) or pactlitaxel 90 mg/m2 weekly x 3 of a 28 day cycle (Regimen B) followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3-6: 30 min) every 21 days x 6 cycles. Maintenance bevacizumab (MB) started after the completion of combination of paclitaxel and bevacizumab and it was given at a dose of 15 mg/kg intravenously once every 21 days for a maximum of 8 cycles. Patients were allowed to receive growth factors. Dose reductions were done based on hematologic and non-hematologic toxicities.

ELIGIBILITY:
INCLUSION CRITERIA

* Baseline measurements and evaluations must be obtained within 4 weeks of registration to the study. Abnormal PET scans will not constitute evaluable disease, unless verified by computed tomography (CT) scan or other appropriate imaging
* At least 1 objective measurable disease parameter by Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Unresectable locally advanced or metastatic angiosarcoma
* ≤ 2 prior chemotherapeutic regimens for angiosarcoma
* No prior paclitaxel, docetaxel, or bevacizumab for angiosarcoma (previous paclitaxel or docetaxel allowed if not given for angiosarcoma and more than 12 months has elapsed since last dose)
* No evidence of other active malignancies other than carcinomas in-situ of the cervix or basal cell carcinoma of the skin within 6 months prior to registration
* If history of deep venous thrombosis or pulmonary embolism, receiving a stable dose of anticoagulation therapy for at least 2 weeks prior to registration
* Within 7 days prior to registration, use of any anti-platelet drugs, such as ticlopidine, clopidogrel, and cilostazol. The use of aspirin or other nonsteroidal anti-inflammatory drugs (NSAID) is allowed
* ECOG performance status 0 to 2
* Patients must have adequate organ function as evidenced by the following laboratory studies (within 2 weeks prior to registration):
* Serum creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 x upper limit of normal (ULN). If documented hepatic involvement, can be ≤ 3 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) or Aspartate aminotransferase (AST) < 2 x ULN. If documented hepatic involvement, can be ≤ 5 x ULN
* Absolute neutrophil count ≥ 1500/mm3 and platelet count > 100,000/mm3
* Platelets ≤ 1.5 x ULN
* International normalized ratio (INR) ≤ 1.5 x ULN
* Partial thromboplastin time (PTT) ≤ 1.5 x ULN
* Left ventricular ejection fraction ≥ 50%
* ≥ 18 years
* Women of childbearing potential must have a negative human chorionic gonadotropin (hCG) pregnancy test within 2 weeks prior to registration

EXCLUSION CRITERIA

* Life expectancy < 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an another experimental drug study
* Inadequately-controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known central nervous system (CNS) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Significant vascular disease (eg, aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a urine protein: creatinine ratio (UPC) ratio ≥ 1.0 at screening
* Known hypersensitivity to any component of bevacizumab
* Active infection requiring parental antibiotics
* Known human immunodeficiency virus (HIV) infection
* Pregnant or breast feeding
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2016-03 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N Ganjoo, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Santa Monica Sarcoma Center, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - MD Anderson Sarcoma Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A Treatment 1: Participants were to receive paclitaxel 200 mg/m² intravenously over 3 hours every 21 days followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3 to 6: 30 min) every 21 days x 6 cycles.
  Maintenance bevacizumab (MB), 15 mg/kg once every 21 days intravenously for a maximum of 8 cycles, was initiated after the completion of paclitaxel + bevacizumab combination.
- Regimen B Treatment 2: Patients were to receive paclitaxel 90 mg/m² weekly x 3 of a 28-day cycle followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3 to 6: 30 min) every 21 days x 6 cycles.
  Maintenance bevacizumab (MB), 15 mg/kg once every 21 days intravenously for a maximum of 8 cycles, was initiated after the completion of paclitaxel + bevacizumab combination.
Period: Screening
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Started | 9 | 9
Completed | 8 | 8
Not Completed | 1 | 1
Not completed — Screen Failure | 1 | 1
Period: Treatment Cycles 1 to 3
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Started | 8 | 8
Completed | 6 | 5
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Discontinued, < 3 cycles treatment | 2 | 2
Period: Inter-treatment Period
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Started | 6 | 5
Completed | 6 | 2
Not Completed | 0 | 3
Not completed — Did not start Cycle 4 | 0 | 3
Period: Treatment Cycles 4 to 6
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The primary objective of this study was to evaluate progression-free survival (PFS or non-progression rate) through 4 months from start of treatment.
  Progression is defined as ≥ 20% increase in the sum of the longest diameter of target lesions, as compared to the baseline measurements, and/or the appearance of one or more new lesion(s).
Time Frame: 4 months
Population: Includes all subjects that started treatment
Measure: Number; unit: Participants without disease progression
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Number analyzed (Participants) | 8 | 8
Participants without disease progression | 4 | 5

2. Secondary Outcome: Overall Response Rate After 3 Cycles
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria, per protocol. Overall response rate (ORR) is the sum of the Complete Response (CR) + Partial Response (PR) rates. The ORR for participants after 3 cycles of treatment (12 weeks) is expressed as the number and proportion of subjects.
  RECIST Criteria
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s),
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: 12 weeks
Population: Includes participants that complete 3 cycles of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Number analyzed (Participants) | 6 | 5
Participants
  Complete Response (CR) | 1 | 0
  Partial Response (PR) | 2 | 2
  Stable Disease (SD) | 1 | 2
  Progressive Disease (PD) | 2 | 1

3. Secondary Outcome: Overall Response Rate After 6th Cycle
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria, per protocol. Overall response rate (ORR) is the sum of the Complete Response (CR) + Partial Response (PR) rates. The ORR for participants after 6 cycles of treatment (24 weeks) is expressed as the number and proportion of subjects.
  RECIST Criteria
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s),
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: 6 Cycles
Population: Includes participants that complete 6 cycles of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Regimen A Treatment 1: Patients were to receive paclitaxel (A) 200 mg/m² intravenously over 3 hours every 21 days followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3-6: 30 min) every 21 days x 6 cycles. Maintenance bevacizumab (MB) started after the completion of a combination of paclitaxel and bevacizumab and it was given at a dose of 15 mg/kg intravenously once every 21 days for a maximum of 8 cycles.
- Regimen B Treatment 2: Patients were to receive paclitaxel (B) 90 mg/m² weekly x 3 of a 28 day cycle followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3-6: 30 min) every 21 days x 6 cycles. Maintenance bevacizumab (MB) started after the completion of a combination of paclitaxel and bevacizumab and it was given at a dose of 15 mg/kg intravenously once every 21 days for a maximum of 8 cycles.
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
Number analyzed (Participants) | 6 | 2
Participants
  Complete Response (CR) | 1 | 0
  Partial Response (PR) | 2 | 0
  Stable Disease (SD) | 1 | 1
  Progressive Disease (PD) | 2 | 1

4. Secondary Outcome: Overall Survival (OS) at 6 Months
Description: Assessed as the number of subjects known to remain alive 6 months after study entry
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Regimen A / Treatment 1: Participants were to receive paclitaxel 200 mg/m² intravenously over 3 hours every 21 days followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3 to 6: 30 min) every 21 days x 6 cycles.
  Maintenance bevacizumab (MB), 15 mg/kg once every 21 days intravenously for a maximum of 8 cycles, was initiated after the completion of paclitaxel + bevacizumab combination.
  Bevacizumab: 15 mg/kg, IV every 21 days x 6 cycles.
  Paclitaxel: Regimen A / Treatment 1: 200 mg/m² IV over 3 hours every 21 days.
  Regimen B / Treatment 2: 90 mg/m² weekly x 3 of a 28-day cycle
- Regimen B / Treatment 2: Patients were to receive paclitaxel 90 mg/m² weekly x 3 of a 28-day cycle followed by bevacizumab 15 mg/kg intravenously over (cycle 1: 90 min; cycle 2: 60 min; cycles 3 to 6: 30 min) every 21 days x 6 cycles.
  Maintenance bevacizumab (MB), 15 mg/kg once every 21 days intravenously for a maximum of 8 cycles, was initiated after the completion of paclitaxel + bevacizumab combination.
  Bevacizumab: 15 mg/kg, IV every 21 days x 6 cycles.
  Paclitaxel: Regimen A / Treatment 1: 200 mg/m² IV over 3 hours every 21 days.
  Regimen B / Treatment 2: 90 mg/m² weekly x 3 of a 28-day cycle
Arm/Group | Regimen A / Treatment 1 | Regimen B / Treatment 2
Number analyzed (Participants) | 8 | 8
Participants | 7 | 8

5. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: Assessed as the number of subjects known to remain alive 12 months after study entry
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A / Treatment 1 | Regimen B / Treatment 2
Number analyzed (Participants) | 8 | 8
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | Regimen A Treatment 1 | Regimen B Treatment 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 8/8 | 4/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A Treatment 1 (N=8) | Regimen B Treatment 2 (N=8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Increased right hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mechanical fall
Fever (General disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Colon perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Circumflex artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Progression of aggressive tumor (General disorders) | 1 (1) | 0 (0)
Pleuritic right chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A Treatment 1 (N=8) | Regimen B Treatment 2 (N=8)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intermittent nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intermittent vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intermittent diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intermittent stomach pain/ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Occasional indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Occasional abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gas pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia intermittent (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Worsening pain left flank (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth sores (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth irritation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ateration in taste (Gastrointestinal disorders) | 0 (0) | 2 (2)
Metallic taste (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 4 (6) | 4 (5)
Headache (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 3 (3) | 0 (0)
Intermittent fever (General disorders) | 0 (0) | 1 (1)
Worsened hypertension (Vascular disorders) | 1 (1) | 0 (0)
Intermittent dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Restless legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Worsening peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy feet (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy toes (Nervous system disorders) | 3 (3) | 0 (0)
Numbness/tingling feet (Nervous system disorders) | 1 (1) | 0 (0)
Numbness/tingling hands (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy fingertips (Nervous system disorders) | 2 (2) | 2 (2)
Sensory neuropathy fingers/toes (Nervous system disorders) | 1 (1) | 0 (0)
Intermittent xerostomia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sensory neuropathy both lower extremities (Nervous system disorders) | 0 (0) | 1 (1)
Tingling fingertips (Nervous system disorders) | 0 (0) | 1 (1)
Pain left leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
occasional pain on left scalp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain left face (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Worsened R hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia intermittent (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Epistaxis intermittent (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Delerium (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 4 (4) | 7 (7)
Thrombocytopenia (Investigations) | 3 (8) | 0 (0)
Elevated alkaline phosphatase (Investigations) | 3 (8) | 1 (1)
Elevated Aspartate Aminotransferase (Investigations) | 1 (1) | 2 (2)
Elevated Alanine Aminotransferease (Investigations) | 1 (2) | 1 (4)
Hyperbilirubinemia (Investigations) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated uric acid (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated potassium (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Prolonged international normalized ratio (Investigations) | 1 (1) | 0 (0)
Increased creatinine (Investigations) | 1 (1) | 0 (0)
Increased B-natriuretic peptide (Investigations) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnea-Occasional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increasing shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Easy bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gait disorder (General disorders) | 2 (2) | 0 (0)
Hot flashes occasional (General disorders) | 1 (1) | 0 (0)
Bilateral crackles lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 2 (3) | 0 (0)
Pain-Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Change in vision (Eye disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Difficulty walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — from fall
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pruritus nontargert lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash on extremites (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash chest (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash back of neck (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Nail infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin peeling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cold intolerance (General disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased oral cavity bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Voice changes (General disorders) | 2 (2) | 0 (0)
Edema left arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Earache (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Scalp tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Afebrile neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Edema Left hand (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema left knee (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache-occasional (General disorders) | 1 (1) | 1 (1)
Hemoglobinemia (Blood and lymphatic system disorders) | 3 (10) | 2 (3)
Hyperpigmented macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — on tips of fingers/toes
Intermittent fever (Infections and infestations) | 1 (1) | 0 (0)
Intermittent leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic pain feet (Nervous system disorders) | 1 (1) | 0 (0)
Night sweats (Nervous system disorders) | 1 (1) | 0 (0)
Nose hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain left chest wall- occasional (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Worsened anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Numbness tingling toes/soles (Nervous system disorders) | 1 (1) | 0 (0)
Rash arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Occasional hypertension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pain right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Occasional diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Occasional headache (Nervous system disorders) | 0 (0) | 1 (1)
Occasional nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Occasional Hypomagnesemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Occasional hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Oral irritation (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No